CLINICAL TRIAL: NCT01422850
Title: A Prospective, Open Phase I Study to Investigate the Tolerability and Efficacy of Administering Repeated Doses of ALECSAT to Prostate Cancer Patients.
Brief Title: Safety Study of Repeated Dosing of a Cytotoxic Lymphocytes (CTL) Based Prostate Cancer Therapy
Acronym: ALECSAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CytoVac A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV002
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Hormone-refractory Prostate Cancer
Keywords: hormone-refractory prostate cancer; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: ALECSAT — Autologous activated CTL and NK-cells injected as three intravenous injections interspaced by 5 weeks.

SUMMARY:
This study is a phase I study of a cell based prostate cancer therapy, Autologous Lymphoid Effector Cells Specific Against Tumor-cells (ALECSAT). Safety and tolerability of a single dose has been shown in 13 prostate cancer patients. In this study 20 prostate cancer patients will receive 3 doses of the ALECSAT treatment. In this therapy specific cells from the patient's own immune system are isolated, activated and re-administered to the patient to boost a specific immune response against the cancer cells. The aim of the study is to show safety and tolerability for repeated dosing of this type of therapy. It is the hypothesis that the cells administered during the therapy will attack the tumor cells and in this way stop or slow down the progression of disease.

DETAILED DESCRIPTION:
This study is a prospective open phase I study to investigate the safety and tolerability of administration of repeated doses of a cell based medicinal product (CBMP) ALECSAT.

ALECSAT is an autologous CBMP that is made from the patient's own blood cells. ALECSAT contains a large amount of tumour specific cytotoxic Lymphocytes (CTL) and Natural Killer (NK) cells that are isolated activated and amplified in number.

The CBMP is given as a slow i. v. injection to patients with prostate cancer. The patients are in the late stage of the disease where they have received hormone treatment but their disease is progressing.

The primary objective of the study is to observe if any side effects or tolerability issues occur as a consequence of the repeated administration of ALECSAT, secondarily it will be observed if changes in Prostate-Specific Antigen (PSA) levels or any positive anti tumor effect may be observed. The study has the purpose to investigate whether repeated treatment with ALECSAT in any way is toxic.

Trial Design: The study is an open, prospective phase I safety study of ALECSAT in prostate cancer patients.

A group consisting of 4 patients will be treated twice with ALECSAT according to the protocol. Then an interim analysis will be done. If there are no signs of significant toxicity related to the treatment, the study will continue to the third treatment for these patients and with 14 more patients that will be treated with ALECSAT according to the protocol. Thus this study will include a total of 20 patients.

The patients will after the first administration of ALECSAT be hospitalized for 2 days. Five and 10 weeks later the patients will be hospitalized for 1 day and receive the second and third administration of ALECSAT. Each patient will furthermore be followed closely for 12 weeks after the third treatment. During the course of the entire study the patients will be monitored by 11 planned study visits, by the investigators at Department of Urology, Fredrikssund Hospital, Denmark.

ELIGIBILITY:
Inclusion Criteria:

1. Serum castration levels of testosterone, (total testosterone under 1.7nmol/l).
2. Three consecutive rises of PSA minimum 1 week apart, resulting in at least two 50 % increases over the PSA nadir.
3. Antiandrogen withdrawal for at least 4 weeks, or PSA progression despite secondary hormonal manipulations, or progression of osseous or soft tissue lesions.
4. Be over the age of 18 and capable of understanding the information and giving informed consent.
5. Expected survival time (life expectancy) of over 6 months.
6. Adequate performance status better than 2 (WHO/ECOG Performance status score).

Exclusion Criteria:

1. A low blood count (haemoglobin < 6.0 mmol/l).
2. Lymphocyte counts below 0.8 x 109/l.
3. Positive tests for anti-HIV-1/2; HBsAg, anti-HBc (Hepatitis B Core Antigen) and Anti-HCV (Hepatitis C Virus).
4. Syphilis i.e. being positive in a Treponema Pallidum test.
5. Uncontrolled serious bacterial, viral, fungal or parasitic infection.
6. Clinically significant autoimmune disorders or conditions of immune suppression.
7. Treatment with corticosteroids (steroid hormones) or bisphosphonates or have been in chemotherapy or radiation treatment one month prior to inclusion in the clinical trial.
8. Blood transfusions within 48 hours prior to donation of blood for ALECSAT production.
9. Inclusion in other clinical trials 6 weeks prior to inclusion in the trial or enrolment in other clinical trials during the ALECSAT clinical trial.
10. Any medical condition that will render participation in the study risky or, according to the Investigator will make the assessment of side effects difficult.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Meyhoff, MD, Principal Investigator — Department of Urology, Frederikssund Hospital, Frederikssundsvej 30, 3600 Frederikssund
Locations (1):
- Department of Urology, Frederikssund, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects was recruited consecutively. The subjects were hospitalized on the day ALECSAT was administered and also one day after the first administration. The overall study period for each participating patient was 25 weeks. The subjects were followed closely during 12 weeks after last treatment by planned study visits.
Groups:
- ALECSAT: After inclusion in the ALECSAT trial, the subject donates 200 ml blood sample for the first ALECSAT product, and after 6 and 11 weeks the subject donated 200 ml again for the second and third product. ALECSAT was thereafter administered at week 4, 9, and week 14.
Period: Overall Study
Arm/Group | ALECSAT
Started | 21
Week 4 - First Treatment | 21
Week 5 | 20 (One patient withdrawn by PI due to progressive disease)
Week 9 - Second Treatment | 20
Week 14 - Third Treatment | 19 (One patient withdrawn by PI and referred to external radiotherapy due to progressive disease.)
Week 15 | 18 (One patient withdrawn by PI due to increased PSA. Started bicalutamide treatment.)
Completed | 18
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | ALECSAT
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years]
  Mean age | 71 [56 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  Denmark | 21

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: To show safety and tolerability patients was monitored closely after administration of ALECSAT and during the follow up period. Heart rate, temperature, blood pressure, Performance status was monitored. Blood samples analysed were: PSA, Alkaline Phosphatase (ALP), Lactate DeHydogenase (LDH), Creatinine (CREAT) and Standard haematology: Blood picture (complete blood count, haemogram), leucocytes, Differential count, electrolytes, renal function, and liver count (liver enzymes).
  AE and SAE was reported during the study period and the Investigator was urged to judge whether the event was related to the study product or not.
Time Frame: At planned study visit´s at study week 0, 4, 5, 6, 7, 9, 10, 11, 12, 14, 15, 16, 18, 21, 24 and at study visit week 25
Population: No formal statistical analysis plan was considered for this study. Any subject that received one administration of ALECSAT and a 6 week follow-up period will be considered as having received ALECSAT and be included in the efficacy part of the report. All patients that received at least one injection of ALECSAT was assessed for safety.
Measure: Number; unit: Events
Arm/Group | ALCESAT
Number analyzed (Participants) | 21
Events
  Total numbers of Adverse Events (AE) | 67
  AE judged as related to study product | 8
  Number of Serious Adverse Events (SAE) | 9
  SAE judged as related to study product | 0
  Safety issues identified by EORTC | 0

2. Secondary Outcome: The Secondary Endpoint for This Study is to Establish if Any Indications of a Positive Therapeutic Effect on the Prostate Cancer May be Observed.
Description: No significant conclusion of efficacy is possible due to the study design with only one group of patients. However by analyzing and comparing the outcome with the data the individual patient presented at baseline some trends of efficacy, defined as stable disease or partial response, are possible. Trends towards possible treatment response were measured by monitoring PSA, a potential marker for prostate cancer disease progression; by other blood markers; and by Quality of life questionnaire (EORTC QLQ-C30) and WHO/ECOG (Eastern Cooperative Oncology Group). Control of any bone metastases were followed by hotspots and bone scan index measured by skeletal scintigraphy.
Time Frame: Within 12 weeks
Measure: Number; unit: participants
Groups:
- Trends Towards Possible Treatment Response: No significant conclusion of efficacy is possible due to the study design with only one active group of patients. However by analyzing and comparing the outcome with the data the individual patient presented at baseline some trends of efficacy are possible. Scintigraphy and blood tests (PSA, ALP, LDH and Creatinine)were used for this analysis.
Arm/Group | Trends Towards Possible Treatment Response
Number analyzed (Participants) | 21
participants
  Trends towards possible treatment response | 11
  No trends of possible treatment response | 8
  Not evaluable patients | 2

3. Primary Outcome: Blood Pressure, Pulse and Temperature
Description: Blood pressure, pulse and temperature were monitored frequently during 48 hours post injection of the study product, and thereafter at each follow up visit.
Time Frame: At planned study visit´s at study week 0, 4, 5, 6, 7, 9, 10, 11, 12, 14, 15, 16, 18, 21, 24 and at study visit week 25
Measure: Number; unit: participants
Arm/Group | ALECSAT
Number analyzed (Participants) | 21
participants
  Significant abnormal changes in Blood pressure | 0
  Significant abnormal changes in Pulse | 0
  Significant abnormal changes in temperature | 0

ADVERSE EVENTS:
Time Frame: At planned study visit´s at study week 0, 4, 5, 6, 7, 9, 10, 11, 12, 14, 15, 16, 18, 21, 24 and at study visit week 25
Description: At each visit, the physician must assess whether any adverse events/reactions or side effects have occurred. Such events may either be reported by the subjects, be observed at the visits or discovered by the laboratory tests.
Arm/Group | ALECSAT
Serious Adverse Events (participants affected / at risk) | 7/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALECSAT (N=21)
Back pain radiating to legs (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain in pelvis area radiating to leg. Not associated with the study product.
Increased blood Creatinine (Renal and urinary disorders) | 1 (1) — Hospitalization due to elevated Serum Creatinine. Not associated with the study product.
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Increased thigh pain bilateral. Withdrawn by PI due to skeletal metastasis. Referred to external radiotherapy. Not associated with the study product.
Ureter obstruction (Renal and urinary disorders) | 1 (1) — Stone in urethra BEFORE first dose of the study product. Not associated with the study product.
General physical health deterioration (General disorders) | 1 (1) — Shortness of breath and blurred vision. Thorax scanning verifies vertebral metastasis in the lung level. Withdrawn from the study due to progressive disease. Not associated with the study product.
Femoral artery bypass (Vascular disorders) | 1 (1) — Femoral bypass due to thrombosis. Not associated with the study product.
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Fracture due to accidental fall. Not associated with the study product.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Elective surgery/excision of malignant melanoma performed at three times due to node metastasis. Not associated with the study product.
Paroysmal atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALECSAT (N=21)
Allergic conjunctivitis (Eye disorders) | 1 (1)
Noose bleed (Vascular disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 3 (3)
Warm but no fever (General disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hydronephros (Renal and urinary disorders) | 1 (1)
Flu (General disorders) | 1 (1)
Lip sore/cold (Skin and subcutaneous tissue disorders) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 2 (2)
Pain (General disorders) | 11 (16)
Tiredness (General disorders) | 3 (4)
Traumatic injury (Musculoskeletal and connective tissue disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred visison (Eye disorders) | 2 (2)
Cold (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Gout (Renal and urinary disorders) | 1 (1)
Increased creatinine level (Renal and urinary disorders) | 1 (1)
Knee surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Elective knee surgery
Malignant melanom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) — elective surgery; removal of glandulae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less